CLINICAL TRIAL: NCT06759415
Title: Investigation of the Effects of Proprioceptive Neuromuscular Facilitation Techniques and Core Stabilization Exercises on Physical and Functional Parameters in Adolescents With Idiopathic Scoliosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kirsehir Ahi Evran Universitesi (Other)
Responsible Party: Principal Investigator, Mehmet Hanifi Kaya, Pilot Project Manager Lecturer Doctor., Kirsehir Ahi Evran Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 55485
Record Dates: First submitted 2024-06-05; First posted 2025-01-06 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Adolescent Idiopathic Scoliosis
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to either the PNF group or the core stabilization group using a computer-generated randomization list to ensure equal distribution of participants across the two groups.
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor did not know which group the participants were in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PNF group (Active Comparator): Proprioceptive Neuromuscular Facilitation Group: The Proprioceptive Neuromuscular Facilitation (PNF) PNF exercises focused on enhancing neuromuscular control, flexibility, and strength of the spinal and core muscles. The exercise regimen included spiral and diagonal movement patterns, rhythmic stabilization, and contract-relax techniques. Participants were instructed on the activation of the transverse abdominus (TrA) muscle, starting with palpation techniques to feel the muscle contraction. Exercises progressed from supine positions to more challenging postures, incorporating breathing control to avoid the Valsalva maneuver.
  Interventions: Other: Exercise
- core stabilization group (Active Comparator): Core Stabilization Group: The core stabilization exercises aimed to improve the stability and strength of the core muscles, which are crucial for maintaining spinal alignment and posture. The exercise regimen included static and dynamic postural control exercises, balance training, and functional movement patterns. The core stabilization exercises focused on strengthening the deep trunk muscles, including the transverse abdominis, multifidus, and pelvic floor muscles.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Exercise therapy was applied to individuals in both groups.

SUMMARY:
Adolescent Idiopathic Scoliosis (AIS) is a prevalent three-dimensional torsional disorder, primarily affecting adolescents during puberty. Characterized by a lateral deviation of the spine greater than 10°, AIS can lead to physical and psychological issues, including back pain, cosmetic deformity, and reduced quality of life. This study aims to compare the effects of Proprioceptive Neuromuscular Facilitation (PNF) techniques and Core Stabilization exercises on physical and functional parameters in adolescents with idiopathic scoliosis. This randomized controlled trial was conducted with 52 adolescents aged 10-18 years, diagnosed with AIS (Cobb angle of 10-30°). Participants were randomly assigned to either the PNF group or the Core Stabilization group. Both groups underwent a 10-week supervised exercise program, supplemented by a home exercise regimen. Primary outcomes included changes in the Cobb angle and Angle of Trunk Rotation (ATR). Secondary outcomes assessed quality of life (SRS-22), perceived trunk appearance (WRVAS), and physical function (6MWT and STS).

DETAILED DESCRIPTION:
Adolescent Idiopathic Scoliosis (AIS) is a prevalent three-dimensional torsional disorder, primarily affecting adolescents during puberty. Characterized by a lateral deviation of the spine greater than 10°, AIS can lead to physical and psychological issues, including back pain, cosmetic deformity, and reduced quality of life. This study aims to compare the effects of Proprioceptive Neuromuscular Facilitation (PNF) techniques and Core Stabilization exercises on physical and functional parameters in adolescents with idiopathic scoliosis. This randomized controlled trial was conducted with 52 adolescents aged 10-18 years, diagnosed with AIS (Cobb angle of 10-30°). Participants were randomly assigned to either the PNF group or the Core Stabilization group. Both groups underwent a 10-week supervised exercise program, supplemented by a home exercise regimen. Primary outcomes included changes in the Cobb angle and Angle of Trunk Rotation (ATR). Secondary outcomes assessed quality of life (SRS-22), perceived trunk appearance (WRVAS), and physical function (6MWT and STS).

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 10 and 18 years old,
2. First-time diagnosis of AIS,
3. Risser sign of 0-3 and a Cobb angle of 10-30°,
4. Sanders classification of 0-6,
5. Lenke curve Type 1 or Type 1A,
6. Volunteered to participate in the study.

Exclusion Criteria:

1. The presence of other types of scoliosis (e.g., congenital or neuromuscular scoliosis),
2. a history of spinal surgery,
3. use of a brace,
4. contraindications for exercise (e.g., cardiovascular or respiratory disorders),
5. previous AIS treatment,
6. rheumatological diseases, and/or other neuromuscular problems.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 52 (Actual)
Dates: Start 2022-01-12 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2023-02-10 (Actual)

PRIMARY OUTCOMES:
Cobb | 24 weeks
  The Cobb: Lines are drawn parallel to the upper edge of the superior vertebra and the lower edge of the inferior vertebra. Then, perpendicular lines are drawn to these parallel lines, and the angle between the two perpendiculars is measured. This angle, known as the Cobb angle, indicates the degree of scoliosis.

SECONDARY OUTCOMES:
The Walter Reed Visual Assessment Scale | 24 weeks
  WRVAS: Perceived trunk appearance was evaluated using the Walter Reed Visual Assessment Scale (WRVAS), which assesses the cosmetic impact of scoliosis from the patient's perspective. The WRVAS consists of seven items, each scored from 1 (no deformity) to 5 (severe deformity), with a higher total score indicating a greater perceived deformity.
Trunk Rotation Angle, | 24 weeks
  Trunk Rotation Angle: The ATR was evaluated using a scoliometer and Adam's forward bend test. Participants were asked to bend forward, and the ATR was measured at the apical vertebrae of the curve. This measurement is sensitive to changes in the rotational aspect of the scoliosis deformity.
Scoliosis Research Society-22 | 24 weeks
  Scoliosis Research Society-22: Quality of Life was assessed using the Scoliosis Research Society-22 (SRS-22) questionnaire, a validated self-report instrument that measures health-related QoL across five domains: function/activity, pain, self-image/appearance, mental health, and satisfaction with management. The total score is the average of the domain scores.

CONTACTS AND LOCATIONS:
Locations (1):
- Mehmet Hanifi KAYA, Kırşehir, Kırşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No